CLINICAL TRIAL: NCT00002265
Title: An Open-Label, Multicenter Study to Evaluate the Safety and Tolerability of Dideoxycytidine (ddC) in Patients With AIDS or Advanced ARC Who Previously Demonstrated Intolerance to Zidovudine (AZT) in Protocol N3300 or N3492
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 031C; N3526A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1994-02

CONDITIONS: HIV Infections
Keywords: Zalcitabine; Drug Evaluation; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zalcitabine

INTERVENTIONS:
Drug: Zalcitabine

SUMMARY:
To demonstrate that zalcitabine (dideoxycytidine; ddC) monotherapy is safe and tolerable in the treatment of patients with AIDS or advanced AIDS related complex (ARC) who previously demonstrated intolerance to zidovudine (AZT) treatment while in Protocol N3300 (NIAID ACTG 114) or N3492 (NIAID ACTG 119).

NOTE OF CAUTION FOR CONCOMITANT MEDICATIONS ON STUDY:

Patients on amphotericin, pyrimethamine, sulfadiazine, trimethoprim/sulfamethoxazole, ganciclovir, intravenous pentamidine, intravenous acyclovir or oral acyclovir or other bone marrow or renal toxic drugs may not tolerate concomitant ddC. If these drugs are given concomitantly with ddC, patients should have frequent clinical and laboratory assessments, as appropriate. Drugs that are nephrotoxic or have the potential to cause peripheral neuropathy might be expected to cause increased toxicity when co-administered with ddC. Drugs that could cause serious additive toxicity when co-administered with study medication will be allowed for treatment of an acute intercurrent illness or opportunistic infection at the discretion of the investigator. Their use may be allowed with interruption of study drug for up to 35 days per episode, for a total of 90 days for the study. If the patient's condition requires chronic administration of these medications, the patient will be discontinued from study medication and followed.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Recommended:

* Prophylactic aerosolized pentamidine.
* Allowed for maintenance after recovering from infection for which initially prescribed:
* Pyrimethamine.
* Sulfadiazine.
* Amphotericin.
* Fluconazole.
* Ketoconazole (= or < 400 mg/day).
* Acyclovir ( = or < 1000 mg/day).
* Ganciclovir.
* Medications for tuberculosis or Mycobacterium avium infection.
* Allowed:
* Erythropoietin.
* Megace.
* Trimethoprim/sulfamethoxazole < or = 20 mg/kg/day.
* Nystatin.
* Low dose acetaminophen or non-steroidal anti-inflammatory agents ( = or < 3 g/day).
* Medications on which patient has been stable for 14 days prior to study entry.
* Allowed if no evidence of peripheral neuropathy at study entry:
* Isoniazid (must be receiving pyridoxine = or > 50 mg/day concomitantly).
* Phenytoin, if stable for = or > 3 months.
* Metronidazole with a study medication interruption and pre and post testing for peripheral neuropathy. Any signs of this and the patient will not be restarted on study medication.
* REFER TO NOTE OF CAUTION IN PROTOCOL SUMMARY.

Patients must have the following:

* Previously enrolled in NIAID ACTG 114 or NIAID ACTG 119.
* Experienced = or > grade 3 zidovudine (AZT) related toxicity while enrolled in the assigned protocol and followed the procedures for the study drug dose reduction, interruption, rechallenge and permanent discontinuation as per NIAID ACTG 114 or NIAID ACTG 119.
* NOTE:
* After permanent study drug discontinuation from NIAID ACTG 114 the drug code may be broken ONLY after discussion with Hoffmann-La Roche regarding toxicity management and probable relationship to AZT. Although NIAID ACTG 119 is an open-label study, investigators should also contact Hoffmann-La Roche prior to entering any patient into this protocol.
* Toxicities must be "probably" AZT related (as determined by the investigator and following discussion by sponsor) for patients to be eligible for inclusion into this protocol.
* Toxicities must be resolved to = or < grade 2 within 45 days of discontinuation from AZT in NIAID ACTG 114 or NIAID ACTG 119.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* An active AIDS defining opportunistic infection or other active intercurrent illnesses if their ongoing treatment requires the use of excluded medications (see Exclusion - Concurrent Medications).
* Baseline fever > 38.5 C if caused by an occult opportunistic infection or neoplasm and requiring continuous treatment with excluded medications. If the evaluation for infection is unrevealing, the patient may be entered after the evaluation is completed but while mycobacterial cultures are still pending. Patients with a history of unexplained fever > 38.5 C should be evaluated as above and/or be afebrile (T < 38.0 C) for 2 weeks prior to study entry.
* Severe AIDS dementia complex as defined by a score of < 23 on the Mini-Mental State Exam at the time of discontinuation from NIAID ACTG 114 or NIAID ACTG 119.
* Any history of peripheral neuropathy or moderate to severe peripheral neuropathy as defined below:
* A score of = or > 4 in any one category or a score of = or > 2 in two categories of the peripheral neuropathy segment of the Signs and Symptoms Questionnaire.
* Accompanied by:
* Results on the Standardized Neurological exam indicative of a moderate abnormality, particularly impaired sensation of sharp pain, light touch or vibration in lower extremities, distal extremity weakness or distal extremity hyporeflexia.
* Significant cardiac disease, defined as history of ventricular arrhythmias requiring medication, prior myocardial infarct or history of angina or ischemia changes on EKG.
* Significant liver disease, as defined by transaminases > 5 x upper limit of normal or a history of cirrhosis or ascites.
* Significant renal disease as defined by an estimated creatinine clearance < 50 ml/min.

Concurrent Medication:

Excluded:

* Other antiretroviral agents.
* Biologic modifiers.
* Corticosteroids.
* Other experimental agents including:
* Foscarnet.
* Ribavirin.
* ddI.
* Drugs that could cause peripheral neuropathy including:
* Hydralazine.
* Nitrofurantoin.
* Vincristine.
* Cisplatin.
* Dapsone.
* Disulfiram.
* Diethyldithiocarbamate.

Patients with the following are excluded:

* An active AIDS defining opportunistic infection or other active intercurrent illnesses if their ongoing treatment requires the use of excluded medications (see Exclusion - Concurrent Medications). Such patients will be allowed into the study if they have completed therapy with an excluded concomitant medication and are stable for 14 days. Had to discontinue study medication in NIAID ACTG 114 or NIAID ACTG 119 because of an opportunistic infection or intercurrent illness which required continuous treatment with medications allowed for concomitant administration in NIAID ACTG 114 or ACTG 119. Symptoms and conditions defined in patient Exclusion - Co-Existing Condition. Active substance or alcohol abuse. Unwillingness or deemed unable to sign informed consent.

Prior Treatment:

Excluded within 30 days of study entry:

* Radiation therapy.

Active substance or alcohol abuse.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Davies Med Ctr, San Francisco, California
  - Mount Zion Med Ctr, San Francisco, California
  - Ctr for Special Immunology, Fort Lauderdale, Florida
  - Dr Robert Swartz, Fort Myers, Florida
  - Med Service, Miami, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Henry Ford Hosp, Detroit, Michigan
  - Graduate Hosp, Philadelphia, Pennsylvania
  - Humana Hosp / Med City Dallas, Dallas, Texas